CLINICAL TRIAL: NCT04437459
Title: The Reproducibility and Clinical Utility of an Abbreviated Fat Tolerance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: HS1844
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Dyslipidemias; Metabolic Syndrome
MeSH Terms: conditions — Dyslipidemias; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abbreviated Fat Tolerance Test (Experimental)
  Interventions: Other: High-fat shake
- Oral Glucose Tolerance Test (Active Comparator)
  Interventions: Other: Pure glucose solution

INTERVENTIONS:
Other: High-fat shake — Participant consumes a high-fat test shake. Blood is drawn before and 4 hours after this shake to measure triglycerides.
  Arms: Abbreviated Fat Tolerance Test
Other: Pure glucose solution — Participant consumes 75 grams of pure glucose. Blood is drawn before and 2 hours after this drink to measure glucose.
  Arms: Oral Glucose Tolerance Test

SUMMARY:
This study aims to evaluate the reliability of a shortened fat tolerance test ("abbreviated fat tolerance test", or "AFTT") for measuring post-meal lipids in human blood. The reliability of the triglyceride results in this test are compared to the reliability of the glucose results from an oral glucose tolerance test (OGTT), a widely-used and clinically accepted metabolic test.

ELIGIBILITY:
Inclusion Criteria:

* Free of chronic disease
* Normal (healthy) fasting glucose and triglycerides

Exclusion Criteria:

* Presence of pace-maker
* Pregnant
* Using tobacco products
* Using medications or dietary supplements that could modify primary outcomes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Reliability of the Change in Triglycerides after a High-Fat Meal | The two fat tolerance tests are separated by 1 week.
  Participants complete two fat tolerance tests. In each test, triglycerides are measured in blood immediately before and 4 hours after consumption of a high-fat meal. The reliability/agreement in measuring the triglyceride change between the 2 tests is being determined.
Reliability of the Change in Glucose after Ingestion of a Glucose Solution | The two glucose tolerance tests are separated by 1 week.
  Participants complete two glucose tolerance tests. In each test, glucose is measured in blood immediately before and 2 hours after consumption of a pure glucose solution. The reliability/agreement in measuring the glucose change between the 2 tests is being determined.

CONTACTS AND LOCATIONS:
Overall Officials: Sam R Emerson, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States